CLINICAL TRIAL: NCT04722380
Title: Nigella Sativa Oil Extract and Xenograft Bone Graft in Treatment of Infra-bony Defects: a Combined Clinical and Histological Study
Brief Title: Nigella Sativa Oil Extract and Xenograft Bone Graft in Treatment of Infra-bony Defects
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Doaa Ahmed Yousef, lecturer, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2021-01-13; First posted 2021-01-25 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Localized Aggressive Periodontitis
Keywords: Nigella Sativa oil extract; Localized Aggressive Periodontitis

STUDY DESIGN:
Intervention Model Description: 10 patients, twenty sites with, localized aggressive periodontitis, with CAL ≥ 5 will be included in the present study. Sites will be allocated randomly to be surgically treated with, Nigella Sativa oil extract Mixed with xenograft or xenograft alone.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- test group (Experimental): 10 infrabony defects treated surgically with Nigella Sativa oil extract Mixed with xenograft
  Interventions: Procedure: periodontal regenerative surgery
- control group (Placebo Comparator): 10 infrabony defects treated surgically with xenograft alone
  Interventions: Procedure: periodontal regenerative surgery

INTERVENTIONS:
Procedure: periodontal regenerative surgery — Procedure/Surgery: open flap debridement Open flap for removal of diseased periodontal tissues and necrotic cementum , using xenogenic bone graft with or without Nigella Sativa oil extract
  Other Names: periodontal surgery

SUMMARY:
The aim of this study will be to evaluate, clinically, and radiographically the effect of Nigella Sativa oil extract Mixed with xenograft versus xenograft alone in the treatment of intra-bony defects in patients with aggressive periodontitis.

DETAILED DESCRIPTION:
in 10 patients, twenty sites in subjects with, localized aggressive periodontitis, with CAL ≥ 5 will be included in the present study. Sites will be allocated randomly to be surgically treated with, Nigella Sativa oil extract Mixed with xenograft or xenograft alone. At baseline, 3, 6 after surgery, the following clinical parameters (PD, CAL, BOP) and CBCT at baseline and 6 months x-ray will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* systemically healthy patients were selected

  * patients who had not received any medications for the previous six months that may interfere with periodontal tissue health or healing.
  * Patients should demonstrate their ability to maintain good oral hygiene

Exclusion Criteria:

* • Smokers and pregnant patients.

  * Medically compromised patients and systemic conditions precluding periodontal surgery.
  * Subjects who do not comply with oral hygiene measures as evidenced in recall visits.
  * Restoration or caries in the site to be treated or non-vital tooth
  * Restoration or caries in the site to be treated or non-vital tooth

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-11-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
probing pocket depth | 6 months
  probing pocket depth probing pocket depth will be recorded at baseline, 3, and 6 months at the site to be treated
clinical attachment level | 6 months
  clinical attachment level will be recorded at baseline, 3, and 6 months at the site to be treated
bleeding on probing | 6 months
  bleeding on probing will be recorded at baseline, 3, and 6 months at the site to be treated
cone beam x ray measuring bone fill | 6 months
  bone fill will be recorded at baseline, and 6 months at the site to be treated

CONTACTS AND LOCATIONS:
Overall Officials: doaa bayoumi, PHD, Principal Investigator — Tanta University
Locations (1):
- Doaa Ahmed yousef bayoumi, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No